CLINICAL TRIAL: NCT02214017
Title: Can a Telemedicine Strategy With Home Treatment Save Resources in Acute Medical Conditions While Maintaining Quality of Care?
Brief Title: Telemedicine Strategy With Home Treatment Save Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Ole Winther Rasmussen, Senior Consultant, Associate Professor, Kolding Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Telemedicine in type 2 DM
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; telemedicine; glycemia; lipids; blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Diabetic patients attended usual procedure in the outpatient clinic with regular visits
  Interventions: Behavioral: Behavioral motivation
- Telemedicine group (Experimental): After initial check-up in the outpatient dept. medical treatment, control of blood glucose, blood pressure, lipids, and education was executed via videotelephone in the telemedicine group. A videotelephone, TandBerg E20, in the telemedicine group was delivered and serviced by the Danish Tele Company, TDC.
  Interventions: Device: A videotelephone, TandBerg E20,; Behavioral: Behavioral motivation

INTERVENTIONS:
Device: A videotelephone, TandBerg E20,
  Arms: Telemedicine group
Behavioral: Behavioral motivation — Optimization of medical care in diabetes

SUMMARY:
Progress in technology has made telemedicine-based solutions with video consultations available in the management and treatment of chronic diseases like diabetes, heart failure and lung insufficiency at home. However, no direct comparisons on health outcomes of telemedicine using video consultations versus usual outpatient treatment are available.

We wanted to implement a model of telemedicine and to evaluate health indicators in type 2 diabetes patients treated by video consultations or the standard outpatient treatment

DETAILED DESCRIPTION:
Chronic illnesses, such as asthma, diabetes, heart failure, and hypertension, represent a significant burden of disease Chronic diseases also impose huge costs on the health care systems responsible for managing them as well as their significance for those affected.

Non-pharmacological treatment is mandatory for type 2 diabetes patients characterized by central obesity, sedentary lifestyle, and overeating (1). Secondary failure to reach treatment goals despite an extensive National diabetes rehabilitation program in Denmark is often seen (2). Outpatient control shows positive effects on outpatient rehabilitation (3) reducing HbA1c, weight, and blood pressure. However, some patients never accomplish good diabetes regulation and in others regulation deteriorates over time. New approaches are required and need testing to motivate and give feedback to the patients at home. Telemedicine has the capacity to achieve this, where a diabetic nurse may optimize motivation, treatment, and diet through direct feedback adapted to milieu of the patient in accordance with a potential spouse.

Good metabolic control is important as diabetes is inevitable a factor for increased risk of cardiovascular disease, neuropathy, and nephropathy (4). The quality of life and reduction in work ability is affected, thus, life expectancy is shortened by 6-8 years. Multi-factorial intervention may delay this (5).

The high incidence of the serious implications strengthens the importance of achieving good metabolic control through lifestyle changes. Health education shows reduction in cardiovascular risk factors (6-8), which often disappears after the end of the intervention (6-8). Good self-care and compliance improve the outcome and reduces diabetes complications (9) and we need new tools to achieve higher attendance to the National diabetes program. Telemedicine represents a novel tool of educating and controlling chronic diseases. It reduced HbA1c for five years with in trials designed to test video-conferencing, clinical data entry and review, web-based education materials, and monitored chat groups (10). Home telemonitoring was compared with telephone calls reducing the HbA1c levels in type 2 diabetes (11) and the technology confer a statistically significant reduction in HbA1c of 0.5 % when applied as add-on to standard treatment. It was used adjunctively to a broader telemedicine initiative for adults with diabetes. The largest telemedicine study initiated by the Ministry of Health in England (Whole Systems Demonstrator) randomized 3320 patients [12] with heart failure and diabetes to telemedicine care. It showed that the telemedicine intervention as add-on therapy resulted a statistically significant reduction in mortality from 8.3% versus 4.6%. Similarly, it showed a reduction of number of inpatients and the number of bed days by 11% and 14%, respectively. The patients' health-related quality of life was unchanged. The savings was less than the additional cost of using telemedicine and overall it cost 15% more per patient. This point at two important factors when applying telemedicine solutions: First, it should preferably replace the standard care and not add-on and, second, be based on the patient's own computer, tablet or smartphone, all of which will reduce the cost substantially. Telemedicine is available for 98-99% of all inhabitants in Denmark by broadband, which allows video conference at home. A few randomized trials with this technology are available at present. We aimed at implementing a telemedicine model in our setting and the design and method should evaluate the quality of treatment as well as technical problems and replace the standard treatment.

Aim:

We compared clinical data from a telemedicine group with a standard care group treated by the same medical algorithm. We wanted to reduce the barriers for the use of a home monitoring and -treatment among elderly, type 2 diabetes patients

Hypothesis:

Treatment by telemedicine or standard care in type 2 diabetes patients results in similar clinical HbA1c, blood pressure, and lipids.

Materials and methods:

Individually visits at the outpatient clinic to plan improvement of glycemic control were made before information of the study was given. Individual goals of the treatment and the drugs needed to fulfil the objectives were agreed on. The patients received the information for the study, and if they wanted to participate, they signed an approval of participation and randomization was performed. All medical treatment, control of blood glucose, blood pressure, lipids, and education was executed via videotelephone in the telemedicine group In the control group patients attended usual procedure in the outpatient clinic with regular visits. Summary of recommendations for glycemic, blood pressure, and lipid control for the participants were: HbA1c 6.5-7.5% (48-58 mmol/L) , fasting blood glucose 6.5-7.5 mmol/l, diurnal blood pressure < 130/80 mmHg, LDL-cholesterol <100 mg/dL (<2.5 mmol/L) and start of medication with elevated urinary albumin/creatinine excretion ≥30 (μg/mg). The treatment algorithm was lifestyle adjustment plus antidiabetic drugs described elsewhere. When the goals were reached within 3 weeks, the videotelephone was disconnected and patients were encouraged to continue glycemic control at their general practitioner. However, the trial went on with a follow-up and evaluation after six month according to the 'intention-to-treat' principle to see if a difference in the initial care mattered significantly.

A videotelephone in the telemedicine group was delivered and serviced by the Danish Tele Company. The trial included type 2 diabetes patients allocated from October 2011 until July 2012 referred to the outpatient clinic from general practitioners. At entry, all patients were screened by albumin/creatinine excretion rate, blood pressure, and electrocardiogram, lipid profile, diabetic food control, and arteriosclerotic symptoms (angina pectoris, claudication, and fatigue). Diurnal blood pressure was measured by monitors. All measurements were repeated six months after inclusion in all participants

ELIGIBILITY:
Inclusion Criteria:

The participants had to live at home, be able to communicate by videotelephone, had no psychiatric disorders, an age between 40 and 85 years and be able to administer medication. -

Exclusion Criteria:

Exclusion criteria were type 1 diabetes, speech disabilities, non-Danish speakers or with severe chronic disease like renal failure (GFR<30 ml/min), liver insufficiency or in cancer treatment.

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ole W Rasmussen, Dr.Med.Scie, Principal Investigator — Kolding Sygehus
Locations (1):
- Endrinology Dept, Kolding Hospital, Kolding, Denmark

REFERENCES:
- [Background] Bower P, Cartwright M, Hirani SP, Barlow J, Hendy J, Knapp M, Henderson C, Rogers A, Sanders C, Bardsley M, Steventon A, Fitzpatrick R, Doll H, Newman S. A comprehensive evaluation of the impact of telemonitoring in patients with long-term conditions and social care needs: protocol for the whole systems demonstrator cluster randomised trial. BMC Health Serv Res. 2011 Aug 5;11:184. doi: 10.1186/1472-6963-11-184. PMID 21819569
- [Background] Shea S, Weinstock RS, Teresi JA, Palmas W, Starren J, Cimino JJ, Lai AM, Field L, Morin PC, Goland R, Izquierdo RE, Ebner S, Silver S, Petkova E, Kong J, Eimicke JP; IDEATel Consortium. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus: 5 year results of the IDEATel study. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):446-56. doi: 10.1197/jamia.M3157. Epub 2009 Apr 23. PMID 19390093
- [Background] Stone RA, Rao RH, Sevick MA, Cheng C, Hough LJ, Macpherson DS, Franko CM, Anglin RA, Obrosky DS, Derubertis FR. Active care management supported by home telemonitoring in veterans with type 2 diabetes: the DiaTel randomized controlled trial. Diabetes Care. 2010 Mar;33(3):478-84. doi: 10.2337/dc09-1012. Epub 2009 Dec 15. PMID 20009091
- [Background] Wootton R. Twenty years of telemedicine in chronic disease management--an evidence synthesis. J Telemed Telecare. 2012 Jun;18(4):211-20. doi: 10.1258/jtt.2012.120219. PMID 22674020
- [Result] Rasmussen OW, Lauszus FF, Loekke M. Telemedicine compared with standard care in type 2 diabetes mellitus: A randomized trial in an outpatient clinic. J Telemed Telecare. 2016 Sep;22(6):363-8. doi: 10.1177/1357633X15608984. Epub 2015 Oct 14. PMID 26468213
- Available data/document: publication: doi: 10.1177/1357633X15608984 — https://www.ncbi.nlm.nih.gov/pubmed/26468213

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemedicine Group: After initial check-up in the outpatient dept. medical treatment, control of blood glucose, blood pressure, lipids, and education was executed via videotelephone in the telemedicine group. A videotelephone, TandBerg E20, in the telemedicine group was delivered and serviced by the Danish Tele Company, TDC.
  A videotelephone, TandBerg E20,
  Behavioral motivation: Optimization of medical care in diabetes
Period: Overall Study
Arm/Group | Standard Care | Telemedicine Group
Started | 22 | 18
Completed | 22 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Telemedicine Group | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 13 | 6 | 19
Age, Continuous [Median (Full Range); unit: years] | 68 [36 to 80] | 59 [46 to 83] | 64 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 14 | 13 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 22 | 18 | 40
BMI [Median (Full Range); unit: kg / m^2] | 30 [23 to 43] | 32.7 [26 to 67] | 31.8 [23 to 67]
duration of type 2 diabetes [Median (Full Range); unit: years] | 9.5 [0 to 22] | 11.5 [2 to 21] | 11 [0 to 22]
insulin treatment [Count of Participants; unit: Participants] | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Glycemia
Description: Percent of glycosylated hemoglobin, HbA1c
Time Frame: Six months of treatment
Measure: Median (Full Range); unit: percent of glycosylated hemoglobin
Arm/Group | Standard Care | Telemedicine Group
Number analyzed (Participants) | 22 | 18
percent of glycosylated hemoglobin | 7.1 [5.8 to 9.6] | 7.6 [6.2 to 11.9]

2. Secondary Outcome: Lipids
Description: Total-cholesterol
Time Frame: Six months of treatment
Measure: Median (Full Range); unit: milli mols/l
Arm/Group | Standard Care | Telemedicine Group
Number analyzed (Participants) | 22 | 18
milli mols/l | 3.9 [2.7 to 4.9] | 3.6 [2.4 to 4.5]

3. Other Pre Specified Outcome: Blood Pressure
Description: Diurnal blood pressure measured by Spacelab monitor, Spacelab 90207
Time Frame: Six months of treatment
Population: diastolic blood pressure
Measure: Median (Full Range); unit: mmHg
Arm/Group | Standard Care | Telemedicine Group
Number analyzed (Participants) | 22 | 18
mmHg | 73 [50 to 92] | 80 [58 to 95]

ADVERSE EVENTS:
Arm/Group | Standard Care | Telemedicine Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No